CLINICAL TRIAL: NCT02611024
Title: Phase I/II, Multicenter, Open-label, Clinical and Pharmacokinetic Study of Lurbinectedin in Combination With Irinotecan in Pretreated Patients With Selected Advanced Solid Tumors
Brief Title: Pharmacokinetic Study of Lurbinectedin in Combination With Irinotecan in Patients With Selected Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-014-15
Record Dates: First submitted 2015-11-05; First posted 2015-11-20 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors; Glioblastoma; Soft Tissue Sarcoma (Excluding GIST); Endometrial Carcinoma; Epithelial Ovarian Carcinoma; Mesothelioma; Gastroenteropancreatic Neuroendocrine Tumor; SCLC; Gastric Carcinoma; Pancreatic Adenocarcinoma; Colorectal Carcinoma; Neuroendocrine Tumors
Keywords: Lurbinectedin; PM01183; Tumors; Cancer; Pharma Mar; Sarcoma; SCLC; Neuroendocrine
MeSH Terms: conditions — Glioblastoma; Sarcoma; Endometrial Neoplasms; Carcinoma, Ovarian Epithelial; Mesothelioma; Gastro-enteropancreatic neuroendocrine tumor; Stomach Neoplasms; Colorectal Neoplasms; Neuroendocrine Tumors; Neoplasms | interventions — PM 01183; Irinotecan

STUDY DESIGN:
Intervention Model Description: Patients with selected advanced solid tumors will be divided into 3 groups: the Lurbinectedin Escalation Group, the Irinotecan Escalation Group and the Intermediate Escalation group. Each group will have a different dose escalation scheme.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lurbinectedin Escalation Group (Experimental): Irinotecan 75 mg/m^2 as a 90-min (-5-min/+30-min) intravenous (i.v.) infusion, followed by Lurbinectedin with starting dose of 1.0 mg/m^2 as a 60-min (-5-min/+20-min) i.v. infusion followed by Irinotecan alone on Day 8 (at the same dose as Day 1 and as a 90-min [-5-min/+30-min] i.v. infusion)
  Interventions: Drug: Lurbinectedin; Drug: Irinotecan
- Irinotecan Escalation Group (Experimental): Starting dose of Irinotecan 15 mg/m^2 as a 90-min (-5-min/+30-min) i.v. infusion, followed by Lurbinectedin 3.0 mg/m^2 as a 60-min (-5-min/+20-min) i.v. infusion followed by Irinotecan alone on Day 8 (at the same dose as Day 1 and as a 90-min [-5-min/+30-min] i.v. infusion).
  Interventions: Drug: Lurbinectedin; Drug: Irinotecan
- Intermediate Escalation Group (Experimental): Starting dose of Irinotecan 50 mg/m^2 as a 90-min (-5-min/+30-min) i.v. infusion, followed by Lurbinectedin 2.6 mg/m^2 as a 60-min (-5-min/+20-min) i.v. infusion. No Irinotecan dose will be administered on Day 8 in this group.
  Interventions: Drug: Lurbinectedin; Drug: Irinotecan

INTERVENTIONS:
Drug: Lurbinectedin — lurbinectedin (PM01183) 4 mg vials
  Other Names: PM01183
Drug: Irinotecan — irinotecan 40 mg, 100 mg or 300 mg vials

SUMMARY:
Prospective, open-label, dose-ranging, uncontrolled phase I/II study of Lurbinectedin in combination with irinotecan. The study will be divided into two stages: a Phase I dose escalation stage and a Phase II expansion stage.

DETAILED DESCRIPTION:
Phase I dose escalation stage.

During the Phase I escalation stage, patients with selected advanced solid tumors will be divided into three groups: the Lurbinectedin Escalation Group, the Irinotecan Escalation Group and the Intermediate Escalation Group. Each group will have a different dose escalation scheme. A treatment cycle is defined as an interval of three weeks.

Three to six patients will be included at each dose level. If dose-limiting toxicity (DLT) occurs in less than one third of evaluable patients in each cohort, escalation can proceed to the next dose level within each group.

The MTD in each group will be the lowest dose level explored during dose escalation in which one third or more of evaluable patients develops a DLT in Cycle 1. At any dose level, if one among the first three evaluable patients has a DLT, the dose level should be expanded up to six patients. Dose escalation will be terminated once the MTD or the last dose level is reached, whichever occurs first, except if all DLTs occurring at a given dose level are related to neutropenia (i.e., febrile neutropenia, grade 4 neutropenia lasting > 3 days or neutropenic sepsis) in which case dose escalation may be resumed, starting at the same dose level and following the same original schedule but with mandatory primary G-CSF prophylaxis.

Once the MTD has been reached, a minimum of nine evaluable patients will be recruited at the immediately lower dose level (or at the last dose level if the MTD is not defined yet): this level will be confirmed as the RD if less than one third of the first nine evaluable patients develop DLT during Cycle 1.

Phase II expansion stage.

If signs of activity are observed in one or more tumor types, there will be a phase II expansion stage after the RD is defined for each group. A tumor-specific expansion cohort (or cohorts if signs of activity are observed in more than one of the permitted tumor types) at each of these RDs may include approximately 20 treated patients per tumor type. If no indication of efficacy is observed in the dose escalation phase of a specific group, then recruitment of patients into that group may be terminated.

Furthermore, one new cohort of patients with neuroendocrine neoplasms (NENs), with approximately 40 treated patients, will be included in the Phase II expansion stage of this study. Patients in this cohort will be treated at the RD determined during the Phase I escalation stage in the Lurbinectedin Escalation Group (Lurbinectedin 2.0 mg/m2 plus irinotecan 75 mg/m2 with the administration of G-CSF). These patients will be divided into two groups of 20 treated patients each:

* Group 1 will include patients with poorly differentiated grade 3 neuroendocrine cancer (NEC) (Ki67 >20%) of gastroenteropancreatic origin or unknown primary site (excluding lung primary tumors) according to the 2019 World Health Organization (WHO) classification of tumors of the digestive system, after progression to first-line chemotherapy with a platinum-based regimen.
* Group 2 will include patients with well differentiated grade 2 (Ki-67 3-20%) or grade 3 (Ki-67 21-55%) gastroenteropancreatic neuroendocrine tumors (GEP-NETs) according to the 2019 WHO classification of tumors of the digestive system, after progression to no more than three prior lines of systemic therapy.

Following the finding of promising efficacy to date, two expansion cohorts in the Lurbinectedin Escalation Group will be further expanded:

* The cohort of patients with small cell lung cancer (SCLC) will be expanded to at least 100 patients treated in second line.
* The cohort of patients with soft tissue sarcoma (STS) will be expanded with between 25 and 80 treated patients with synovial sarcoma (a subtype of STS)

Only in these two expansion cohorts, an Independent Review Committee (IRC) will determine the response evaluation at each tumor assessment necessary to derive the best patient's response and assign the date of first documentation of response and progression/censoring according to RECIST v.1.1. Operational details for the IRC and the algorithm and its validation by an expert panel are described in detail in the IRC charter.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and dated written informed consent prior to any specific-study procedure.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1.
4. Life expectancy ≥ 3 months.
5. Histologically or cytologically confirmed diagnosis of advanced disease of any of the following tumor types:

   For the Lurbinectedin Escalation Group and the Irinotecan Escalation Group:
   1. Glioblastoma.
   2. Soft-tissue sarcoma (excluding gastrointestinal stromal tumors [GIST]).
   3. Endometrial carcinoma.
   4. Epithelial ovarian carcinoma (including primary peritoneal disease and/or fallopian tube carcinomas and/or endometrial adenocarcinomas) regardless of platinum sensitivity.
   5. Mesothelioma.
   6. Gastroenteropancreatic neuroendocrine tumors (GEP-NET).
   7. Small cell lung cancer (SCLC).
   8. Pancreatic adenocarcinoma.
   9. Gastric carcinoma.
   10. Colorectal carcinoma (CRC).

   For the Intermediate Escalation Group:
   1. Endometrial carcinoma.
   2. SCLC.
   3. Other solid tumors may be included, if appropriate, after discussion between the Investigators and the Sponsor.

   For the Phase II expansion stage:
   1. Glioblastoma.
   2. Soft tissue sarcoma (including synovial sarcoma),
   3. Endometrial carcinoma.
   4. SCLC.
   5. Neuroendocrine tumors.

      * Group 1: Poorly differentiated grade 3 NEC (Ki-67 >20%) according to the 2019 WHO classification of tumors of the digestive system, of gastroenteropancreatic origin or unknown primary site (lung primary tumors will be excluded).
      * Group 2: Well differentiated grade 2 (Ki-67 3-20%) or grade 3 (Ki-67 21-55%) GEP-NETs according to the 2019 WHO classification of tumors of the digestive system.
6. The number of prior lines of therapy allowed per patient will be as follows:

   For the Phase I Escalation Stage:

   No more than two prior lines of cytotoxic-containing chemotherapy regimens for advanced disease

   For the Phase II Lurbinectedin Expansion Stage:
   * For SCLC, one prior line of platinum-containing chemotherapy with/without antibodies against programmed cell death protein-1 (PD-1) or programmed death ligand-1 (PD-L1).
   * For NENs,

     * In Group 1 (patients with poorly differentiated NEC of gastroenteropancreatic origin or unknown primary site, excluding lung primary tumors), one prior line of platinum-based chemotherapy; and
     * In Group 2 (patients with well differentiated GEP-NETs), no more than three prior lines of systemic therapy (that may include somatostatin analogues, chemotherapy, everolimus and/or sunitinib).
   * For all other tumor types, no more than two prior lines of cytotoxic-containing chemotherapy regimens for advanced disease.

   There is no limit for prior targeted therapy, hormonal therapy and immunotherapy (such as nivolumab).
7. Phase II expansion stage: Tumor-specific cohort(s) at the RD:

   1. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1. For patients with glioblastoma: Measurable disease according to RECIST v.1.1 and Response Assessment in Neuro-Oncology (RANO) criteria.
   2. Documented disease progression per RECIST v.1.1 during or immediately after last therapy according to any of the aforementioned criteria. For patients with glioblastoma: Documented disease progression per RECIST v.1.1 and RANO criteria.
8. At least three weeks since the last anticancer therapy, (including immunotherapy, investigational drugs and radiotherapy), and at least six weeks since nitrosoureas and mitomycin C (systemic).

   For biological/investigational anticancer therapies given orally, the aforementioned period of at least three weeks could be changed for one of at least five half-lives (whichever occurred first), provided that the therapy is given as single agent and not combined with other drugs. If this is not the case, this exception will not be acceptable.

   For patients with glioblastoma: at least 12 weeks since the end of radiotherapy, except if:
   1. The patient has a new lesion outside of the radiotherapy field, or
   2. The patient has undergone brain surgery to remove the tumor before study entry, and progressive disease has been confirmed histologically.

   Note: washout periods will be referred to the day of first cycle administration (Day 1), not to the day of registration (Day 0).
9. Adequate bone marrow, renal, hepatic, and metabolic function (assessed ≤ 7 days before inclusion in the trial):

   1. Platelet count ≥ 100 × 10^9/L, hemoglobin ≥ 9.0 g/dL and absolute neutrophil count (ANC) ≥ 2.0 × 10^9/L.
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × the upper limit of normal (ULN), even in the presence of liver metastases.
   3. Alkaline phosphatase (ALP) ≤ 2.5 × ULN (≤ 5 × ULN if disease-related/in the case of liver metastases).
   4. Total bilirubin ≤ 1.5 × ULN or direct bilirubin ≤ ULN.
   5. International Normalized Ratio (INR) < 1.5 (except if patient is on oral anticoagulation therapy).
   6. Calculated creatinine clearance (CrCL) ≥ 30 mL/minute (using Cockcroft-Gault formula).
   7. Creatine phosphokinase (CPK) ≤ 2.5 × ULN.
   8. Albumin ≥ 3.0 g/dL*
10. Recovery to grade ≤ 1 or to baseline from any adverse event (AE) derived from previous treatment (excluding alopecia and/or cutaneous toxicity and/or peripheral neuropathy and/or fatigue grade ≤ 2).

    * Albumin transfusion to increase the blood level in order to fulfill the inclusion criterion is strictly forbidden.

Exclusion Criteria:

1. Concomitant diseases/conditions:

   1. History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular heart disease within the previous year.
   2. Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment.
   3. Myopathy or any clinical situation that causes significant and persistent elevation of CPK (> 2.5 × ULN in two different determinations performed one week apart).
   4. Ongoing chronic alcohol consumption or cirrhosis with Child-Pugh score B or C. Known Gilbert disease.
   5. Active uncontrolled infection.
   6. Known human immunodeficiency virus (HIV) or known hepatitis C virus (HCV) infection or active hepatitis B.
   7. Any past or present chronic inflammatory colon and/or liver disease, past intestinal obstruction, pseudo or sub-occlusion or paralysis.
   8. Evident symptomatic pulmonary fibrosis or interstitial pneumonitis, pleural or cardiac effusion rapidly increasing and/or necessitating prompt local treatment within seven days.
   9. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study
   10. Active Coronavirus disease (COVID-19).
   11. Hypersensitivity to any of the study drugs or their excipients.
2. Prior treatment with lurbinectedin, trabectedin (Yondelis®) or topoisomerase I inhibitors (irinotecan, topotecan, etc.). Prior topoisomerase inhibitors (e.g., irinotecan) are only allowed in patients with colorectal carcinoma or NENs.
3. Prior bone marrow or stem cell transplantation, or radiation therapy in more than 35% of bone marrow.
4. Known brain metastases or leptomeningeal disease involvement. Glioblastoma lesions (primary or locally advanced) are eligible. Exception: patients with brain metastases are eligible provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment (patients taking steroids in the process of already being tapered within two weeks prior to screening are allowed). Brain CT-scan or MRI results must be provided at baseline.
5. Women who are pregnant or breast feeding and fertile patients (men and women) who are not using an effective method of contraception. Women of childbearing potential (WOCBP) must agree to use an effective contraception method to avoid pregnancy during the course of the trial (and for at least six months after the last infusion). Fertile male patients must agree to refrain from fathering a child or donating sperm during the trial and for four months after the last infusion.
6. Limitation of the patient's ability to comply with the treatment or follow-up protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 66 months
  The MTD will be the lowest dose level explored during dose escalation which one third or more of evaluable patients develops DLTs in Cycle 1. DLTs are related AEs during Cycle 1 fulfilling at least 1 of the criteria below:
  * Grade 4 neutropenia lasting >3 days
  * Febrile neutropenia of any duration or neutropenic sepsis
  * Grade 4 thrombocytopenia/Grade 3 with clinically bleeding requiring a transfusion
  * Grade 4 ALT/AST increase/Grade 3 lasting >14 days
  * Grade≥2 increased ALT/AST concomitantly with total bilirubin increase ≥2.0×ULN and normal ALP
  * Grade≥3 diarrhea lasting >5 days and despite adequate corrective treatment
  * Grade≥3 CPK increase
  * Grade≥3 non-hematological related AE, excluding nausea/vomiting, hypersensitivity reactions, extravasations, grade 3 fatigue lasting <1 week and nonclinically biochemical abnormalities
  * Administration delay of Cycle 2 >15 days from the Day 22 due to any related AEs
  * Failure to meet the Day-8 continuation criteria for irinotecan in Cycle 1
Recommended Dose (RD) | 66 months
  The RD will be the highest dose level explored during dose escalation in which fewer than one third of patients develop DLTs during Cycle 1. DLTs are related AEs during Cycle 1 fulfilling at least 1 of the criteria below:
  * Grade 4 neutropenia lasting >3 days
  * Febrile neutropenia of any duration or neutropenic sepsis
  * Grade 4 thrombocytopenia/Grade 3 with clinically bleeding requiring a transfusion
  * Grade 4 ALT/AST increase/Grade 3 lasting >14 days
  * Grade≥2 increased ALT/AST concomitantly with total bilirubin increase ≥2.0×ULN and normal ALP
  * Grade≥3 diarrhea lasting >5 days and despite adequate corrective treatment
  * Grade≥3 CPK increase
  * Grade≥3 non-hematological related AE, excluding nausea/vomiting, hypersensitivity reactions, extravasations, grade 3 fatigue lasting <1 week and nonclinically biochemical abnormalities
  * Administration delay of Cycle 2 >15 days from the Day 22 due to any related AEs
  * Failure to meet the Day-8 continuation criteria for irinotecan in Cycle 1
Response Rate | At least six weeks after treatment initiation, up to 66 months
  Phase II Expansion Stage: Efficacy Response rate is a percentage of patients with any response: partial response or complete response.
  Antitumor activity will be measured according to RECIST v.1.1.
  * An increase of ≥20% from the baseline or new lesion appears represents progressive disease.
  * A decrease in the sum of target disease of ≥30% represents partial response.
  * Stable disease lies between partial response and progressive disease.
  * Complete response is the disappearance of all lesions with nodes measuring <10 mm and normal tumour markers
  Patients included in the tumor-specific expansion cohort(s) at the RD for each group, and in the new cohort of patients with NENs, must be evaluable per RECIST v.1.1 (including ovarian cancer patients). Specifically, patients with glioblastoma must be evaluated per RECIST v.1.1 and RANO criteria. A patient evaluable for efficacy should have received at least one complete dose of lurbinectedin and irinotecan.

SECONDARY OUTCOMES:
Safety evaluation | Since start of the treatment until 30 days after the last administration of study treatment; or until start of a new antitumor therapy or death
  AEs will be graded according to the NCI-CTCAE v.4.
Peak Plasma Concentration (Cmax) | 66 months
  Pharmacokinetic Outcome Measures
Area under the plasma concentration versus time curve (AUC) | 66 months
  Pharmacokinetic Outcome Measures
Volume of distribution based on the terminal half-life (Vz) | 66 months
  Pharmacokinetic Outcome Measures
Volume of distribution at steady state (Vss) | 66 months
  Pharmacokinetic Outcome Measures
Clearance (CL) | 66 months
  Pharmacokinetic Outcome Measures
Half-life (t1/2) | 66 months
  Pharmacokinetic Outcome Measures
Duration of response | Time from date when response criteria are fulfilled to the first date when progression disease, recurrence or death, until 18 months after the inclusion of the last evaluable patient in the study (end of study), whichever occurs
  Evaluable and measurable as per RECIST v.1.1 or RANO for Glioblastoma patients
Progression-free Survival | From the date of first infusion of study treatment to the date of progression or death or until 18 months after the inclusion of the last evaluable patient in the study (end of study), whichever occurs first.
  Time from the date of first infusion of study treatment to the date of progression or death (due to any cause). If progression or death has not occurred at the time of the analysis, the Progression-free Survival (PFS) will be censored on the date of last tumor evaluation.
Overall Survival | From the date of first infusion of study treatment to the date or death or until 18 months after the inclusion of the last evaluable patient in the study (end of study), whichever occurs first.
  Time from the date of first infusion of study treatment to the date of death (due to any cause). Patients with no documented death will be censored at the last date they are known to be alive.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (4):
  - Sarcoma Oncology Center, Santa Monica, California
  - Massachusetts General Hospital -, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Helios Kilinikum Bad Saarow, Bad Saarow
  - Helios Klinikum Berlin Buch, Berlin
- Italy (2):
  - Campus Biomedico, Roma
  - IRCCS Fondazione Candiolo (Turin), Torino
- Spain (12):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Univeristari Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen Del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Inselspital Bern - Medizinische Onkologie, Bern, Switzerland

REFERENCES:
- [Derived] Falcon A, Ponce S, Cote GM, Gil A, Lin JJ, Bockorny B, Martinez J, Kahatt C, Martinez S, Zubiaur P, Siguero M, Cullell-Young M, Jimenez J, Zugazagoitia J, Paz-Ares L. Phase I results on the efficacy, safety and pharmacokinetics of lurbinectedin and irinotecan in advanced solid tumors. Invest New Drugs. 2025 Aug;43(4):955-967. doi: 10.1007/s10637-025-01583-y. Epub 2025 Sep 18. PMID 40963055